CLINICAL TRIAL: NCT03294421
Title: Combined Access Closed Tympanomastoidectomy: Microsurgery Allied to Endoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 50571215.0.0000.5327
Record Dates: First submitted 2017-09-08; First posted 2017-09-27 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Cholesteatoma; Chronic Otitis Media
MeSH Terms: conditions — Cholesteatoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard closed tympanomastoidectomy (Active Comparator): In this group it will be performed the standard technique for closed tympanomastoidectomy, in which a surgical microscope is used.
  Interventions: Procedure: standard closed tympanomastoidectomy
- combined access tympanomastoidectomy (Experimental): In this group a closed tympanomastoidectomy with combined access will be performed. This technique combines the use of a surgical microscope with a rigid endoscope measuring 14cm of length with 0º and 30º angulation.
  Interventions: Procedure: combined access tympanomastoidectomy

INTERVENTIONS:
Procedure: combined access tympanomastoidectomy — Trans canal surgery with the use of a surgical microscope with a rigid endoscope measuring 14cm of length with 0º and 30º angulation allowing better visualization and removal of the cholesteatoma before mastoid debridement. In this surgery, mastoid debridement is conducted only if there was no full endoscopic removal of the cholesteatoma. The other procedures of this type of surgery are similar to the standard tympanomastoidectomy technique.
  Arms: combined access tympanomastoidectomy
Procedure: standard closed tympanomastoidectomy — 1. Supine position and general anesthesia with orotracheal intubation
  2. Antisepsis and placing of sterile fields
  3. Local anesthesia of the external auditory canal with lidocaine 2% and adrenaline 1:100. 000 UI
  4. Retroauricular incision
  5. Removal of the temporal muscle fascia
  6. Elevation of the surgical flap of the tympanic meatus
  7. Visualization and exploration of the cholesteatoma
  8. Exploration of the ossicular chain
  9. Mastoid debridement
  10. Conservation of the upper posterior wall of the auditory conduct
  11. Removal of the cholesteatoma
  12. Tympanoplasty with the temporal fascia
  13. Retroauricular suture with vycril 3.0 and mononylon 4.0
  Arms: standard closed tympanomastoidectomy

SUMMARY:
Chronic otitis media is a prevalent medical condition, leading to important impact in the lives of the individuals with this condition, and a great amount of patients may need surgical intervention. The main objectives of the surgery in these cases are to restore the anatomy of the middle ear, to improve hearing and to remove the infection to avoid further complications. Still, chronic otitis media with cholesteatoma presents high rates of recurrence and residual symptoms after surgery.

The standard technique used for treatment of chronic otitis media is microsurgery. Nonetheless, with the development of new technologies that use endoscopy, it is now possible to use endoscopic surgery to improve the visualization of the cholesteatoma and ear structures by combining both techniques.

This study will evaluate the efficacy of the combined access surgery technique, which is microsurgery combined with endoscopy, for closed tympanomastoidectomy in patients with cholesteatoma. Furthermore, the study aims to compare the results of the combined access technique and the standard technique by randomizing the patients in two groups: one group will receive tympanomastoidectomy by standard technique and the other group will receive combined technique.

DETAILED DESCRIPTION:
Patients with cholesteatoma and medical indication of closed tympanomastoidectomy will be randomized into two groups. In the first group, microsurgical tympanomastoidectomy will be performed; while combined technique will be performed in the other group. The combined technique improves the visualization of the middle ear canal and the mastoid. Herewith, the best visualization of the surgical site facilitates the full removal of the cholesteatoma. In addition to that, the combined technique is less invasive than the standard one, since less bone debridement is required to access the surgical site.

The outcomes of the study will be evaluated through follow up medical appointments and exams. The patients will be followed by monthly medical appointments with otoscopic evaluations for diagnose of possible recurrence of the disease or residual cholesteatoma. Also, audiometry exams will be performed in the third, sixth and twelfth months. Image exams such as nuclear magnetic resonance may be performed at the end of this period to evaluate relapse of the disease if the otoscopic evaluation is inconclusive.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cholesteatoma with indication for closed tympanomastoidectomy.

Exclusion Criteria:

* Patients with malformation of the temporal bone or previous surgery in the ear eligible for the study.

Ages: 5 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2017-09-22 (Actual); Primary Completion 2020-05-07 (Actual); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Recurrence of cholesteatoma. | 12 months post intervention.
  Recurrence of cholesteatoma, which is defined as development of new disease in the same ear (not related with the previous cholesteatoma), will be evaluated through second look surgery or nuclear magnetic resonance.
Residual cholesteatoma | 12 months post intervention.
  Presence of residual cholesteatoma, which is defined as disease that was not fully removed in the first intervention, will be evaluated through second look surgery or nuclear magnetic resonance.

SECONDARY OUTCOMES:
Hearing outcomes | 3 months post intervention.
  Hearing outcomes will be measured through audiometry exams (parameters that will be analyzed in the exam: Pure tone average (PTA) 500.000 Hz to 2.000 Hz and air bone gap) after three months after surgery and compared with the audiometry exam made before the surgery.
Hearing outcomes | 6 months post intervention.
  Hearing outcomes will be measured through audiometry exams (parameters that will be analyzed in the exam: PTA 500.000 Hz to 2.000 Hz and air bone gap) after six months after surgery and compared with the audiometry exam made before the surgery and the audiometry exam made three months after surgery.
Hearing outcomes | 12 months post intervention.
  Hearing outcomes will be measured through audiometry exams (parameters that will be analyzed in the exam: PTA 500.000 Hz to 2.000 Hz and air bone gap) after twelve months after surgery and compared with the audiometry exam made before the surgery and the audiometry exams made three and six months after surgery.
Length of procedure | measured in minutes from the surgical incision until the suture of the skin.
  Compares the length of the closed tympanomastoidectomy with standard technique and the combined access tympanomastoidectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Sady S Da costa, Principal Investigator — Hospital de Clínicas de Porto Alegre; Mauricio LS Da silva, Principal Investigator — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de clínicas de porto alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paparella MM. Current concepts in otitis media. Henry Ford Hosp Med J. 1983;31(1):30-6. No abstract available. PMID 6863004
- [Background] Ghaffar S, Ikram M, Zia S, Raza A. Incorporating the endoscope into middle ear surgery. Ear Nose Throat J. 2006 Sep;85(9):593-6. PMID 17044426
- [Background] Lima Tde O, Araujo TF, Soares LC, Testa JR. The impact of endoscopy on the treatment of cholesteatomas. Braz J Otorhinolaryngol. 2013 Aug;79(4):505-11. doi: 10.5935/1808-8694.20130090. PMID 23929154
- [Background] Badr-El-Dine M, James AL, Panetti G, Marchioni D, Presutti L, Nogueira JF. Instrumentation and technologies in endoscopic ear surgery. Otolaryngol Clin North Am. 2013 Apr;46(2):211-25. doi: 10.1016/j.otc.2012.10.005. PMID 23566907
- [Background] Marchioni D, Soloperto D, Rubini A, Villari D, Genovese E, Artioli F, Presutti L. Endoscopic exclusive transcanal approach to the tympanic cavity cholesteatoma in pediatric patients: our experience. Int J Pediatr Otorhinolaryngol. 2015 Mar;79(3):316-22. doi: 10.1016/j.ijporl.2014.12.008. Epub 2015 Jan 7. PMID 25631934